CLINICAL TRIAL: NCT04663867
Title: Safety and Effectiveness Study of the AngioSafe Peripheral CTO Crossing System
Brief Title: AngioSafe Peripheral CTO Crossing System Study (RESTOR-1 Study)
Acronym: RESTOR-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AngioSafe, Inc. (Industry)
Collaborators: Veranex, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0071
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Artery Occlusion; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AngioSafe Peripheral CTO Crossing System Procedure (Experimental): Use of AngioSafe Peripheral CTO Crossing System to facilitate the intraluminal placement of guidewires beyond Chronic Total Occlusions (CTOs) in the peripheral vasculature.
  Interventions: Device: AngioSafe Peripheral CTO Crossing System

INTERVENTIONS:
Device: AngioSafe Peripheral CTO Crossing System — The AngioSafe Peripheral CTO Crossing System is intended to facilitate the intraluminal placement of guidewires beyond stenotic lesions, including chronic total occlusions (CTOs) in the peripheral vasculature.

SUMMARY:
The study is designed to evaluate the safety and efficacy of the AngioSafe Peripheral CTO Crossing System.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate the safety and effectiveness of the AngioSafe Peripheral CTO Crossing System. The system facilitates the crossing of chronic total occlusions (CTOs) in the peripheral arteries of lower limbs. A minimum of 70 subjects will be treated across selected study enters within the U.S. and followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with protocol requirements and sign informed consent form
* ≥ 22 years of age
* Peripheral arterial disease defined by Rutherford Clinical Classification (Category 2-5)
* Peripheral artery disease in target extremity is confirmed by imaging (catheter angiography, computed tomographic angiography (CTA), and/or magnetic resonance angiography (MRA))

Angiographic Inclusion Criteria:

* Target lesion in native de novo common femoral artery (CFA), superficial femoral artery (SFA), and/or popliteal artery
* Vessel diameter(s) for target lesion is ≥ 3.0mm and ≤ 10mm
* Subject's target lesion is a severely stenosed segment of ≤ 300 mm that involves the CTO(s)
* Subject's target lesion involves at least one CTO that is 99-100% stenosed
* Subject has at least one vessel with run-off to the foot

Exclusion Criteria:

* Systemic infection or an infection in extremity of target lesion
* Target lesion within native vein or synthetic vessel grafts or in stent occlusion
* Planned intervention in the contralateral limb during the study
* Planned intervention in the target limb of the inflow vessels during the study
* Planned intervention of lower extremities after study procedure within 30-day follow-up visit
* Coagulopathy or bleeding diatheses, thrombocytopenia with platelet count less than 50,000/μl, or INR > 1.7
* Antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated
* Allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated
* Allergy to nickel, titanium, urethane, nylon, or silicone
* History of myocardial infarction within 30 days prior to enrollment/consent
* History of stroke within 30 days prior to enrollment/consent
* Chronic kidney disease (CKD) of stage 4 or greater based on an Estimated Glomerular Filtration Rate (eGFR) <30ml/Min, unless the subject is on chronic renal replacement therapy
* Hemoglobin levels <10g/dL verified by a lab test no older than 14 days prior to enrollment, unless the subject has a history of chronic anemia at a stable level, no recent bleeding diathesis or history of blood transfusion in the last six weeks
* Pregnant or nursing, for females of child-bearing potential (< 50 years of age)
* Participating in another interventional research study that may interfere with study endpoints
* Prior major amputation (above ankle) in target extremity
* Acute limb ischemia (ALI)
* Prior unsuccessful attempt to cross the target lesion
* Subject has had a procedure on the target limb or contralateral limb within 7 days
* Subject has had a procedure on the target limb or contralateral limb within the past 30 days and is unstable

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — North Texas Veterans Healthcare System
Locations (18):
- United States (18):
  - Dignity Health - Chandler Regional Medical Center, Chandler, Arizona
  - Adventist Health St. Helena, St. Helena, California
  - Vascular Care Connecticut, Darien, Connecticut
  - Palm Vascular Centers, Miami Beach, Florida
  - Coastal Vascular & Interventional, PLLC, Pensacola, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Vascular Care Group, Wellesley, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - American Endovascular & Amputation Prevention, West Orange, New Jersey
  - Vascular Solutions of North Carolina, Cary, North Carolina
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont Cardiology Services, Kingsport, Tennessee
  - VA North Texas Medical Center, Dallas, Texas
  - Baylor Scott & White, The Heart Hospital Plano, Plano, Texas
  - Cardiovascular Associated of East Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled a total of 79 participants, with only 74 participants analyzed for effectiveness Outcome Measures. Study results (Outcome Measures) are reported for the 74 participants in the "Full Analysis Set (FAS)" Group described below. The 5 excluded participants are described in in other study Groups, excluded from effectiveness analyses, but included in the safety analyses (Adverse Event reporting).
Groups:
- Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures: The Full Analysis Set (FAS) (n=74) includes all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version. These study participants are also included in the safety analysis of all (n=79) study participants.
- Excluded Participants: Earlier Iteration of the Investigational Device: N=4 study participants were excluded from the effectiveness analysis because they were enrolled under a prior version of the Study Protocol and treated with an earlier iteration of the investigational device, whose use was discontinued early on in the study. These study participants are included in the safety analysis of all (n=79) study participants.
- Excluded Participant: Roll-In Subject: N=1 study participant was excluded from the effectiveness analysis because they were enrolled as a "roll-in" subject under a prior version of the Study Protocol. This study participant is included in the safety analysis of all (n=79) study participants.
Period: Overall Study
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures | Excluded Participants: Earlier Iteration of the Investigational Device | Excluded Participant: Roll-In Subject
Started | 74 | 4 | 1
Completed | 74 | 4 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) (n=74) includes all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version. The FAS population is the primary analysis population defined in the Study Protocol and is the only population with reported Baseline Characteristics analysis as pre-specified in the study Statistical Analysis Plan (SAP).
Groups:
- Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures: The Full Analysis Set (FAS) (n=74) includes all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version.
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Hispanic | 8
  Hispanic | 3
  Other, non-Hispanic | 1
  White, non-Hispanic | 61
  Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 74
Arterial Access Type [Count of Participants; unit: Participants] — Population: Twelve (12) participants had Secondary Arterial Access.
  Participants
    Primary Access: Retrograde Femoral | 62
    Primary Access: Antegrade Femoral | 12
    Primary Access: Pedal | 0
    Primary Access: Popliteal | 0
    Secondary Access: number analyzed (Participants) | 12
    Secondary Access: Retrograde Femoral | 1
    Secondary Access: Antegrade Femoral | 2
    Secondary Access: Pedal | 9
    Secondary Access: Popliteal | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success of AngioSafe Peripheral CTO Crossing System
Description: Clinical Success is defined as the ability of the catheter to facilitate placement of a guidewire into the distal lumen in the absence of device-related major adverse events through discharge or 24-hours post-procedure, whichever is sooner.
Time Frame: 24 Hours
Population: The Full Analysis Set (FAS) (n=74) includes all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
Participants | 65

2. Secondary Outcome: Technical Success of AngioSafe Peripheral CTO Crossing System
Description: Technical Success is defined as the ability of the catheter to facilitate placement of a guidewire into the distal lumen.
Time Frame: Procedure, evaluated directly after performing the investigational procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
Participants | 65

3. Secondary Outcome: Procedural Success of AngioSafe Peripheral CTO Crossing System
Description: Procedural Success is defined as the ability of the catheter to facilitate placement of a guidewire into the distal lumen without a procedural complication within 30 days after the procedure. Procedural complication is defined as the need for open or repeat endovascular surgical repair in the treated limb, or a major bleeding event.
Time Frame: 30 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set (FAS): The Full Analysis Set (FAS) (n=74) includes all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version.
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 74
Participants | 65

4. Secondary Outcome: Evaluation of Intraluminal CTO Crossing Facilitated by the Peripheral CTO Crossing System, as Assessed by an Intravascular Ultrasound (IVUS).
Description: Post-procedure IVUS evaluation of Technical Success cases to determine if crossing was performed intraluminally.
Time Frame: Procedure, evaluated directly after performing the investigational procedure
Population: Post-procedure IVUS evaluations were available for only 55 study participants from the Full Analysis Set (FAS) (n=74) of all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 55
Participants
  Total Intraluminal | 44
  Partial Intraluminal with ≥50% of IVUS image frames Intraplaque | 7
  Partial Intraluminal with <50% of IVUS image frames Intraplaque or Extraluminal | 3
  Not Evaluable | 1

5. Secondary Outcome: The Primary Endpoint (Clinical Success) in the Subgroups by the Degree of Calcification (None/Focal/Mild, and Moderate/Severe).
Description: Clinical Success is defined as the ability of the catheter to facilitate placement of a guidewire into the distal lumen in the absence of device-related major adverse events through discharge or 24-hours post-procedure, whichever is sooner, analyzed by degree of calcification in two subgroups: None/Focal/Mild calcification, or Moderate/Severe calcification.
Time Frame: 24-hours
Population: The Full Analysis Set (FAS) (n=74) of all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version included 53 subjects with Moderate to Severe Calcification and 21 subjects with None to Mild Calcification
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
Participants
  Moderate to Severe Calcification: number analyzed (Participants) | 53
  Moderate to Severe Calcification: Clinical Success | 46
  Moderate to Severe Calcification: Failure | 7
  None to Mild Calcification: number analyzed (Participants) | 21
  None to Mild Calcification: Clinical Success | 19
  None to Mild Calcification: Failure | 2

6. Other Pre Specified Outcome: Lesion Crossing Time, Mean
Description: Lesion crossing time is defined as time starting from the placement of the Peripheral CTO Crossing System at the proximal cap to the time the guidewire is placed in the distal true vessel lumen.
Time Frame: Procedure, evaluated during the investigational procedure
Population: Lesion crossing time was available for only 64 study participants from the Full Analysis Set (FAS) (n=74) of all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version.
Measure: Mean (Standard Error); unit: min
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 64
min | 25 (4)

7. Other Pre Specified Outcome: Lesion Crossing Time, Median
Description: as for outcome 6
Time Frame: Procedure, evaluated during the investigational procedure
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: min
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 64
min | 9 [6 to 16]

8. Other Pre Specified Outcome: Rutherford Clinical Classification (RCC) Assessment
Description: The mean change in the Rutherford Clinical Classification (RCC) assessment at 30 days versus baseline. The Rutherford Clinical Classification (RCC) Scale identifies three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. The RCC Scale Categories and associated Clinical Descriptions are as follows: 0 - Asymptomatic, 1 - Mild claudication, 2- Moderate claudication, 3 - Severe claudication, 4 - Ischemic rest pain, 5 - Minor tissue loss, 6 - Ulceration or gangrene.
Time Frame: Baseline, 30-days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: RCC Scores on a scale
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
RCC Scores on a scale
  Mean change in RCC Score | -2.14 (0.17)
  Mean RCC Score at Baseline | 3.40 (0.09)
  Mean RCC Score at 30-Days | 1.25 (0.20)

9. Post Hoc Outcome: Post-CTO-Crossing Track Dimensions: Width
Description: Angiographic images were post-processed and analyzed to demonstrate angiographic visibility of intraplaque channel formation and to quantify the track width.
Time Frame: Procedure, evaluated directly after performing the investigational procedure
Population: The Full Analysis Set (FAS) (n=74) of all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version included n=55 participants with Technical Success (Outcome Measure 2), with angiographic imaging available for n=43 study participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 43
mm | 2.87 (0.74)

10. Post Hoc Outcome: Post-CTO-Crossing Track Dimensions: Diameter
Description: Intravascular Ultrasounds (IVUS) images were post-processed and analyzed to demonstrate IVUS-confirmation of intraplaque channel formation and to quantify the track diameter.
Time Frame: Procedure, evaluated directly after performing the investigational procedure
Population: The Full Analysis Set (FAS) (n=74) of all study participants analyzed for effectiveness with reported Outcome Measures under the final Study Protocol version included n=55 participants with Technical Success (Outcome Measure 2), with IVUS imaging available for n=44 study participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 44
mm | 2.78 (0.73)

11. Post Hoc Outcome: Post-CTO-Crossing Track Dimensions: Cross Sectional Area
Description: Intravascular Ultrasounds (IVUS) images were post-processed and analyzed to demonstrate IVUS-confirmation of intraplaque channel formation, and to quantify the track dimensions.
Time Frame: Procedure, evaluated directly after performing the investigational procedure
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 44
mm^2 | 6.71 (3.7)

12. Other Pre Specified Outcome: Pain Numeric Rating Scale (NRS) Assessment
Description: The mean change in Pain Numeric Rating Scale (NRS) assessment at 30-days versus baseline. The Pain Numeric Rating Scale (Pain NRS) is a unidimensional measure of pain intensity in adults. The NRS is anchored by terms describing pain severity extremes, where 0 represents no pain and 10 represents the worst pain possible. The NRS Ratings and associated Clinical Descriptions are as follows: 0 - No Pain, 1-3 - Mild Pain, 4-6 - Moderate Pain, 7-9 - Severe Pain, 10 - Worst Pain Possible.
Time Frame: Baseline, 30-days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Pain NRS Scores on a scale
Arm/Group | Full Analysis Set (FAS), All Study Participants With Reported Outcome Measures
Number analyzed (Participants) | 74
Pain NRS Scores on a scale
  Mean change in Pain NRS Rating | -3.17 (0.39)
  Mean Pain NRS Rating at Baseline | 5.24 (0.36)
  Mean Pain NRS Rating at 30-days | 2.06 (0.33)

ADVERSE EVENTS:
Time Frame: 30-days
Description: AEs are reported for all study participants (n=79) including the primary analysis population (Full Analysis Set (FAS, n=74), participants enrolled under a prior version of the Study Protocol and treated with an earlier iteration of the device (n=4), and a participant enrolled as a "roll-in" subject under a prior version of the Study Protocol (n=1). Combined AE reporting for all 79 study participants was pre-specified in the study Statistical Analysis Plan (SAP).
Groups:
- All Study Participants: All study participants (n=79), including: n=74 participants treated the investigational device under the final Study Protocol version, n=4 participants enrolled under a prior version of the Study Protocol and treated with an earlier iteration of the investigational device, and n=1 participant enrolled as a "roll-in" subject under a prior version of the Study Protocol, are included in safety analysis of Adverse Events.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 1/79
Serious Adverse Events (participants affected / at risk) | 5/79
Other Adverse Events (participants affected / at risk) | 39/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=79)
Ansel sheath complication (Surgical and medical procedures) | 1
Anemia (Blood and lymphatic system disorders) | 1
Balloon failure (Surgical and medical procedures) | 1
Death (General disorders) | 1 — Death reported 3 days after the investigational procedure. Classified as not related to the investigational device or procedure. The cause of death was listed as "Hypertensive and Atherosclerotic Cardiovascular Disease" on the death certificate.
Hypertension (Cardiac disorders) | 1
Infection (Infections and infestations) | 1
Pain (General disorders) | 1
Pseudoaneurysm (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=79)
Acute digital ischemia (General disorders) | 1
Arterial blush (Vascular disorders) | 1
Arterial dissection (Surgical and medical procedures) | 12
Arterial perforation (Surgical and medical procedures) | 4
Arteriovenous fistula (Vascular disorders) | 1
Bradycardia (Cardiac disorders) | 2
Rutherford Declines (General disorders) | 2
Edema (General disorders) | 7
Hematoma (General disorders) | 1
Hematuria (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 1
Infection (Infections and infestations) | 2
Major depression (Psychiatric disorders) | 1
Nausea (General disorders) | 1
Pain (General disorders) | 8
Tachycardia (Cardiac disorders) | 1
Total occlusion (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04663867/Prot_SAP_000.pdf